

| Title: | |
|---|---|
| Analysis of marg | inal bone loss in implants placed at the soft tissue-bone tissue level. |
| Researchers: | |
| Main: A | hmed Samir Mabrouk Oraby Elkattan |
| 114411. | miled Summ (vidoroux Oracly Enkattan) |
| Collaborators: | |
| | <ul><li>José López López</li><li>Raúl Ayuso Montero</li></ul> |
| | Xavier Roselló Llabrés |
| | Monica Blázquez |
| Centers: | Hospital Dentistry University of Barcelona (HOUB). |
| | Faculty of Medicine and Health Sciences, Dentistry, University of Barcelona. |
| 2nd version of the | Protocol: July,01, 2022. |

#### **SUMMARY**

The subcrestal placement implant has a positive impact on papilla formation and allows an emergence profile suitable for an aesthetic restoration. Its placement allows the implant-abutment interface to be in a position that contributes to bone remodeling in the neck region of the implant, compared to implants placed at bone level (bone-level, crestal placement). Marginal bone loss from implants placedcrestal or subcrestal has shown conflicting results in recent studies.

### 1.- BACKGROUND OF THE SUBJECT

Dental implants have been introduced as an option for replacing missing teeth, since the initial studies of Professor Per-Ingvar Brånemark in the 1950s, there are multiple studies that support it, including (Andersson B, 1995; Arlin M, 1993; Noack et al, 1999; Jemt T, 2017; The accepted criteria for evaluating implant success were proposed by Albrektsson et al. (Albrektsson et al, 1986), who to identify clinical evidence of successful osseointegration and implant survival, suggested that a marginal bone loss of less than 1.5 mm in the first year and 0.2 mm in the following years, it is acceptable after implant loading (Díaz-Sánchez et al, 2019). Over the past three decades, implant success has been evaluated by survival rates, prosthesis stability, radiographic bone loss, and the absence of infection in the peri-implant soft tissues (Albrektsson et al, 1986; Smith and Zarb 1989; Buser et al, 1990, Albrektsson and Zarb 1998, Misch et al, 2008; The progressive knowledge of patients has increasingly required treatments that offer better aesthetics and comfort, making implantology a demanding field, where obtaining osseointegration or meeting the success criteria of implants highlighted by the lack of pain and infection, absence of radiolucency and mobility and possibility of restoration (Buser et al, in the 1990s). Thus, new parameters have been introduced to evaluate the long-term success of implant restorations. Including health status and natural-looking peri-implant soft tissues, prosthodontic parameters, aesthetics and patient satisfaction. However, osseointegration remains the predominant parameter in implantology (Furhauser et al, 2005; Meijer et al, 2005; Annibali et al, 2009; Belser et al, 2009).

Various authors describe that the position of the implant with respect to the crestal bone is a fundamental factor to preserve the bone in the future (Pontes et al, 2008; Novaes et al, 2009; De Siqueira et al, 2017; Wennerberb et al. al, 2003; Although, regarding this issue there continues to be controversy. Thus, some authors recommend placing the

implant below the crest of the bone (i.e., subcrustal placement). They argue that this position will contribute to the preservation of the mucosa (Pontes et al, 2008), helping to obtain an ideal emergence profile in aesthetic areas (Novaes et al, 2009; Di Siquerira et al, 2017) and preventing the surface of the implant is exposed; at the same time that the presence of mucositis or peri-implantitis is reduced (Wennerberg et, 2003). A possible reason for this could be bacterial colonization of the implant-abutment junction, where an inflammatory infiltrate occurs (Do-Nascimento et al, 2012; Hermann et al, 2000; Broggini et al, 2003). This characteristic, in conjunction with a low oxygen concentration, could create an ideal ecosystem for the proliferation of anaerobic bacteria (Piattelli et al, 2003). On the other hand, it could be speculated that deeper implant placement may correlate with deeper pockets and soft tissue inflammation (Siqueira et al, 2017).

In another order of things, the connection of the implant with the abutment involves microspaces. These microspaces (which facilitate the accumulation of bacteria) can influence peri-implant bone resorption along with other factors such as surgical trauma, the establishment of the biological width, the design of the implant and the position of the implant (Palacios-Garzón et al, 2019; Díaz-Sánchez, et al, 2019; Buser et al., 1990). Studies have shown that this microgap varies between 0 and 135 µm (Dellow et al, 1997; Callan et al, 1998). However, what deserves special attention is that, as in teeth, the biological width is formed around the implants, consisting of a junctional epithelium and connective tissue with an average dimension of approximately 2 mm and 1–1.5 mm. respectively (Berglundh et al, 1991). On the other hand, different risk factors can affect implant lifespan, such as anatomical characteristics, chewing dynamics, and proper implant selection, which are important for long-term prognosis. Today, we know that implants with rough surfaces show a statistically higher survival rate than machined implants at all intervals (Levin et al, 2006).

Maintaining the level of the crestal bone around dental implants is essential for their longterm success and survival (Mei et al, 2017; Al Amri et al, 2017; Marcelo-Machado, et al 2018). Factors that may showcrestal bone resorption in dental implants that affect the survival rate of the dental implant, such as the amount of overload stress (Stoichkov et al, 2018), micromotion (King et al, 2002), location and bacterial infiltration of the implantabutment connection (Blanco et al., 2008; Kozlovsky et al., 2007; Tripodi et al., 2015), periodontal phenotype (Linkevicius et al, 2010), bone density (Hermann et al, 2001; Goiato et al, 2014), trauma surgical (Canullo et al, 2012) and maintenance of oral hygiene (Kozlovsky et al, 20007). In the actulaida, several treatment protocols have been proposed to reduce marginal bone loss around implants (Calvo-Guirado et al, 2015; Vohara et al, 2015; Romanos et al, 2014), including implant placement by below the level of the bony crest (subcrestal placement) (Kutan et al, 2015). Furthermore, the subcrestal implant also has a positive impact on papilla formation and allows for an adequate emergence profile for better aesthetic restoration (Vela-Nebot et al, 2006; Koutouzis et al, 2014). In this placement the implant-abutment interface is in a position that contributes to bone remodeling in the neck region of the implant compared to implants placed at bone level (crestal placement) (Outouzis et al, 2011; Charalampakis et al, 2014). On the other hand,

marginal bone loss from subcrustal implants compared to crests has shown contradictory results in recent studies (Gale et al 2013). Thus, some studies reported similar bone levels for both implant placement techniques (Casagrande et al, 2020). Therefore, we believe it is necessary to continue researching in this field, to make decision-making easier for the clinician.

#### 2-JUSTIFICATION

Various treatment protocols have been proposed to reduce marginal bone loss around implants, including placement of implants below the level of the bone crest (subcrestal placement). The supracrestal implant also has a positive impact on papilla formation and allows an emergence profile suitable for an aesthetic restoration. Allowing the implant-abutment interface to be in a position that contributes to bone remodeling in the implant neck region compared to implants placed at bone level (crestal placement). Marginal bone loss from implants placed bestially/subcrestally has shown conflicting results in recent studies. In this study we intend to evaluate bone loss in 100 Tissue level implants from two different commercial companies: Straumann bone level® with the Bio horizon Tissue level® implant. Buying the data obtained with the existing literature.

#### 3- HYPOTHESIS

# 3.1- Main hypothesis

### **Null hypothesis:**

Two different brands of implants behave in the same way in terms of marginal bone loss, if they are placed based on the indications specified by the manufacturer.

# **Alternative hypothesis:**

Two different brands of implants behave in the same way in terms of marginal bone loss, if they are placed based on the indications specified by the manufacturer.:

#### 3- HYPOTHESIS

#### 3.1- Main hypothesis

<u>Null hypothesis:</u> A brand of implant behaves in the same way in terms of marginal bone loss, if it is placed according to the indications specified by the manufacturer (crestal level or supracestal level).

# **Alternative hypothesis:**

A brand of implant does not behave in the same way in terms of marginal bone loss, if it is placed according to the indications specified by the manufacturer (crestal level or supracestal level).

#### 4-OBJECTIVES

## 4.1 Main objective:

To evaluate marginal bone loss in two different brands of implants placed at the bone level.

### 4.2 Secondary objectives:

- Relationship between marginal bone loss and suprabony soft tissue in mm.
- Relationship between marginal bone loss and ISQ value at the time of implantation.
- Relationship between marginal bone loss and torque (in Newton) at the time of implantation.
- Relationship between marginal bone loss and implant location.
- Relationship between marginal bone loss and the degree of periodontal disease.
- Relationship between marginal bone loss and systemic diseases.
- Relationship between marginal bone loss and smoking

### 5- MATERIAL AND METHOD

# 5.1- Study design

It is a prospective clinical study to compare two implants from two different brands of a similar design for their implantation [tissue level] and to evaluate the marginal bone loss of each dental implant in mm. 96 patients will be analyzed (an expected N of 48 per group, hoping to reach at least 100 implants per arm). See calculation of N in point 5.7.

# 5.2- Study population

The patients will be collected from patients who attend the master's degree in medicine, surgery and Oral Implantology, requesting implant-supported treatment. The study population will consist of patients who require treatment with dental implants, either partially or completely edentulous and who accept their placement and participation in the study.4.2.1 Inclusion / exclusion criteria

### 5.3-Inclusion/exclusion criteria

### Inclusion:

• Patients of both sexes, over 18 years of age, who need dental implant placement for prosthetic rehabilitation. Whether partially or completely in both the maxilla and the mandible.

- Patients with residual alveolar ridge with at least 8 mm of bone height and 4 mm of width.
- Patients must have the ability to understand and decide at the time of voluntarily signing the informed consent before carrying out any intervention related to the study.
- Patients who, after being informed about the objectives and procedures of the research, agree, will sign the informed consent form. And they are ready to carry out the different study visits.

#### **Exclusion:**

- Patients with uncontrolled systemic diseases (ASA  $\geq$  III).
- Patients who do not have 8mm bone height and/or 4mm width
- Patients who require bone regeneration
- Patients with severe periodontal disease or acute pericoronitis.
- Pregnant and breastfeeding women.
- Patients with Deficient or Inadequate Oral Hygiene.
- Patients with severe bruxism.
- Patients taking bisphosphonates or other antiresority medications.
- Smoker of more than 10 cigarettes/day.
- Patients with uncontrolled diabetes mellitus.
- Psychiatric illnesses or unrealistic expectations.
- Immunocompromised or immunosuppressed patient.

# 5.4.-Recruitment

The sample will be for convenience and will be obtained from patients of the Hospital Odontològic Universitat de Barcelona (HOUB) who come to the service of the Master of Dentistry in Oral Medicine, Surgery and Implantology. Once the protocol is approved by the Ethics and Research Committee with Medicines and Health Products of the same HOUB (CEIm-HOUB), the recruitment of study participants will begin, estimated to take one year and 2 months, starting in November 2022.

### 5.5.- Procedures

#### 5.5.1 First session and recruitment

In this first session, before starting surgery and prosthodontic treatment, a thorough medical history will be taken. Each patient will be examined by extra-oral and intra-oral examination, in addition to the evaluation of their respective orthopantomography and cone beam computed tomography (CBCT), to evaluate the level of height and width of the bone for the placement of dental implants. This process will be carried out by the main researcher and supervised by another expert in Dentistry. Study participants who meet the inclusion criteria will then be recruited and asked if they wish to participate. Each of them will be given the following records.

If the patient meets the criteria and is interested, they will sign the informed consent and will be randomized using a randomization table of 10 in 10 implants [e.g.: randomization table ABBAABBAB] to place one type or another of implant:



#### 5.5.2 Second session

The patient will come to the Hospital for primary impressions with alginate. Then a cast will made with gypsum for study the case and bite of the patient will be taken with wax to record it.

#### 5.5.3Third session

The patient will come to the Hospital to operate the surgery within 15-20 days after having the study caste revised by a dentist and specialist from the fixed department. The patient will have temporary prothesis (Fixed or Removable) after the surgery of the implant. A periapical X-Ray will be taken immediately after the surgery to control the marginal bone loss. With the respect to accepted criteria for the assessment of implant success were proposed by Albrektsson and colleagues (Albrektsson *et al.*, 1986), which to identify clinical evidence of successful osseointegration and survival of implants, suggested that a marginal bone loss of less than 1.5 mm in the first year and 0.2 mm in the following years is acceptable after implant loading.

### 5.5.4 Fourth session

Once the osseointegration time has elapsed, 3 months  $\pm$  15 days (in the mandible) and 4 months  $\pm$  15 days (in the maxilla), new clinical and radiographic measurements will be taken and then the rehabilitation phase will begin. The visits will be those corresponding to the required prosthetic treatment (fixed or removable), carried out according to the usual procedures and techniques of the prosthodontic service.

## 5.5.5 Fith session

After placing the prosthesis on the patient, it will be reviewed every 3 months  $\pm$  15 days, for 2 years, to establish controls.

# 5.5.6 Sample's size calculation





Reference points for calculating marginal bone loss. Taken with permission from the author of Lina Dumanova's TFG. Red arrow, known mean of the implant. Green arrows reference the crestal bone and the marginal loss that occurred that allows us to compare at different times of the study.

### 5.6- Description of the treatment or intervention: drugs or techniques to be used.

- All patients will be anesthetized with 2% articaine with epinephrine,
- Regarding medication dispensed:
- Amoxicillin 1000 mg cps /8 hours for 7 days. (Patients allergic to Amoxicilllin, we prescribe Clindamicina 600 mg cps /8H / 7 days).
- Dexketroprofeno 25 mg cps /8 hours for 7 days.
- Omperazol 25 mg cps / 8H/ 7 days for the stomach.
- As rescue medication: Paracetamol 1000 mg cps /8 hours for 7 days and/or Metamizol 650 mg cps 1/8 hours.
- Rinse with 0.12% chlorhexidine 2 times/7 days.

# 5.7.- Sample calculation

According to data obtained in the study by Natalia Palacios-Garzon et al, 2020 (taking into account that both are internally connected implants), in order to detect changes of 0.2mm we would need: Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 48 subjects (implants) in the first group and 48 (Implants) in the second are needed to detect a difference equal to or greater than 0.2 units.

The common standard deviation is assumed to be 0.34. A loss to follow-up rate of 5% has been estimated.

# 5.8.- Statistical analysis

The variable data will be entered into the Excel program of the Microsoft Office 2019 Package (Microsoft Corporation, Washington, USA, 2013) and will be analyzed with the SPSS 26.0 program for Windows (SPSS, Illinois, USA, 2019).

The data collected will be processed using the STATA 14.0 statistical package. A descriptive analysis of the qualitative and quantitative variables will be carried out. The Kolmogorov-Smirnov test will be used to analyze the normality of the measurements.

The relationship between bone loss and implant position will be analyzed using parametric t-test.

The level of statistical significance chosen is 5% ( $\alpha = 0.05$ ). To evaluate the association between the dependent variable bone loss from T0 to T2 and successive Ts and the independent variables implant A, Implant B placement, a multiple linear regression analysis will be used.

All variables considered to potentially affect the study relationship, such as sex, age, and smoking, will be used as control variables in the regression; the number of cigarettes per day, maxilla or mandible, ISQ [implant stability value] and contact of the mesial and distal implant (penseic ade dinets and/or implants by mesial and distal)

#### 5.9- Schedule

| | 2022 | | | | | | | | | 2023 | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | En | Feb | Mar | Abr | May | Jun | Jul | Agos | Sep | Oct | Nov | Dic | En | Feb | Mar | Abr | May | Jun | Jul | Agos | Sep | Oct | Nov | Dic |
| Reclutamiento | | | | | | | | | | | | | | | | | | | | | | | | |
| de | | | | | | | | | | | | | | | | | | | | | | | | |
| participantes | | | | | | | | | | | | | | | | | | | | | | | | |
| | 2024 | | | | | | | | | 2025 | | | | | | | | | | | | | | |
| | En | Feb | Mar | Abr | May | Jun | Jul | Agos | Sep | Oct | Nov | Dic | En | Feb | Mar | Abr | May | Jun | Jul | Agos | Sep | Oct | Nov | Dic |
| Recopilación<br>de datos | | | | | | | | | | | | | | | | | | | | | | | | |
| | En | Feb | Mar | Abr | May | Jun | Jul | Agos | Sep | Oct | Nov | Dic | En | Feb | Mar | Abr | May | Jun | Jul | Agos | Sep | Oct | Nov | Dic |
| Análisis de los<br>datos | | | | | | | | | | | | | | | | | | | | | | | | |

# 5.0- Specification of the acceptance of the national and international ethical norms

The researchers agree that each participating subject will be treated and controlled following the protocol authorized by the Ethics and Research Committee for Medicines and Health Products of the Hospital Odontològic of the University of Barcelona (CEIm-HOUB) and the Declaration of Helsinki of ethical principles for medical research in humans by the World Medical Association (64<sup>a</sup> General Assembly, Fortaleza, Brazil, October 2013).

## 5.1- Economic report

- Cost of rehabilitative prosthetic treatment paid by the patient.
- Administrative costs: in charge of the Master of Dentistry in Medicine surgery and Implant and the doctoral student.
- Material costs: by the Master of Dentistry in Medicine surgery and Implant and the doctoral student.
  - o Ortopantograhia: 31€.
  - o CBCT para un cuadrante: 97€.
  - o CBCT para un mono-implant(Dependente en el caso): 81 €.
  - o Impressional Alginato Aligsul: 10€.
  - o Encerarlo (wax up) GEO CLASSIC gris-OPCA 75GR:20 €.
  - o Dental Gypsum (Snow White plaster): 46€.

- o Implanto Tipo A: 690€.
- o Protesis:830€.
- o Articulado papel (PAPEL BK 01 AZUL 300 HOJAS 0,2mm): 21€.
- o Silicona Optosil P Plus (Heraeus Kulzer GmbH, Hanau, Germany): 80€.
- o Silicona Zetalabor hard 85 shore A (Zhermack, Badia Polesine, Italy): 120€.
- o Guantes de látex (Medicaline, Castellón, España): 180€.

# **5.2- Data collection sheet**

6- BIBLIOGRAPHY

| PERSONAL DATA | |
|---|---|
| CODE: | IN SESSION: |
| NUMBER: | SURNAMES: |
| DATE: | EXAMINER: |
| DATE OF BIRTH (AGE): | SEX: Man□ Woman □ |
| PHONE: | E-MAIL: |
| TYPE OF PATIENT: ASA I ASA II ASA II ASA II PRIMARY DIAGNOSIS (DATE: mm / yyyy | |
| _ | |
| SURGERY TREATMENT (DATE: mm / yy | yy): |
| _ | |
| N° TEETH TO BE REHABILITATED WIT | TH A PROSTHETIC:prosthetic units. |
| TYPE OF PROSTHESIS: | |

- Natalia Palacios-Garzón; Eugenio Velasco-Ortega; José López-López.. Bone Loss in Implants Placed at Subcrestal and Crestal Level: A Systematic Review and Meta-Analysis . Materials (Basel). 2019 Jan 5;12(1):154.Doi: 10.3390/ma12010154.
- María Díaz-Sánchez; María Peñarrocha-DiagO; David Soto-Peñaloza; David Peñarrocha-Oltra.(2019). Influence of supracrestal tissue attachment thickness on radiographic bone level around dental implants: A systematic review and meta-analysis. J Periodontal Res. 2019 Dec;54(6):573-588. Doi: 10.1111/jre.12663. Epub 2019 Jun 23.
- 3. Buser, D.; Weber, H.P.L.N. Tissue integration of non-submerged implants. *Clin. Oral Implants Res.* 1990, *1*, 33–40.
- 4. Mangano, F.; Mangano, C.; Ricci, M.; Sammons, R.L.; Shibli, J.A.; Piattelli, A. Single-tooth Morse taper connection implants placed in fresh extraction sockets of the anterior maxilla: An aesthetic evaluation. *Clin. Oral Implants Res.* 2012, *23*, 1302–1307.
- Donovan, R.; Fetner, A.; Koutouzis, T.; Lundgren, T. Crestal Bone Changes Around Implants With Reduced Abutment Diameter Placed Non-Submerged and at Subcrestal Positions: A 1-Year Radiographic Evaluation. *J. Periodontol.* 2010, 81, 428–434.
- Pontes, A.E.; Ribeiro, F.S.; da Silva, V.C.; Margonar, R.; Piattelli, A.; Cirelli, J.A.; Marcantonio, E., Jr. Clinical and radiographic changes around dental implants inserted in different levels in relation to the crestal bone, under different restoration protocols, in the dog model. *J. Periodontol.* 2008, 79, 486–494.
- 7. Novaes, A.B.; Barros, R.R.M.; Muglia, V.A.; Borges, G.J. Influence of interimplant distances and placement depth on papilla formation and crestal resorption: A clinical and radiographic study in dogs. *J. Oral Implantol.* 2009, *35*, 18–27. [CrossRef] [PubMed]
- 8. De Siqueira, R.A.C.; Fontão, F.N.G.K.; de Sartori IA, M.; Santos, P.G.F.; Bernardes, S.R.; Tiossi, R. Effect of different implant placement depths on crestal bone levels and soft tissue behavior: A randomized clinical trial. *Clin. Oral Implants Res.* 2017, *28*, 1227–1233. [
- 9. Wennerberg, A.; Sennerby, L.; Kultje, C.; Lekholm, U. Some soft tissue characteristics at implant abutments with different surface topography. A study in humans. *J. Clin. Periodontol.* 2003, *30*, 88–94.
- 10. Todescan, F.F.; Pustiglioni, F.E.; Imbronito, A.V.; Albrektsson, T.; Gioso, M. Influence of the microgap in the peri-implant hard and soft tissues: A histomorphometric study in dogs. *Int. J. Oral Maxillofac Implants* 2002, *17*, 467–472.
- 11. Do Nascimento, C.; Miani, P.K.; Pedrazzi, V.; Muller, K.; de Albuquerque Junior, R.F. Bacterial leakage along the implant-abutment interface: Culture and DNA Checkerboard hybridization analyses. *Clin. Oral Implants Res.* 2012, *23*, 1168–1172.
- 12. Hermann, J.S.; Buser, D.; Schenk, R.K.; Cochran, D.L. Crestal Bone Changes Around Titanium Implants. A Histometric Evaluation of Unloaded Non-Submerged and Submerged Implants in the Canine Mandible. *J. Periodontol.* 2000, 71, 1412–1424.
- 13. Broggini, N.; McManus, L.M.; Hermann, J.S.; Medina, R.U.; Oates, T.W.; Schenk, R.K.; Buser, D.; Mellonig, J.T.; Cochran, D.L. Persistent acute inflammation at the implant-abutment interface. *J. Dent. Res.* 2003, *82*, 232–237. [CrossRef] [PubMed]

- 14. Piattelli, A.; Vrespa, G.; Petrone, G.; Iezzi, G.; Annibali, S.; Scarano, A. Role of the Microgap Between Implant and Abutment: A Retrospective Histologic Evaluation in Monkeys. *J. Periodontol.* 2003, 74, 346–352.
- 15. Mina Taheri; Solmaz Akbari; Ahmad Reza Shamshiri; Yadollah Soleimani Shayesteh. (2020). Marginal bone loss around bone-level and tissue-level implants: A systematic review and meta-analysis. 0940-9602/© 2020 Elsevier GmbH. All rights reserved. https://doi.org/10.1016/j.aanat.2020.151525.
- Levin L, Laviv A, Schwartz-Arad D. Long-term success of implants replacing a single molar. J Periodontol. 2006;77:1528–1532.
- 17. Kohen J, Matalon S, Block J, Ormianer Z. Effect of implant insertion and loading protocol on long-term stability and crestal bone loss: A comparative study. J Prosthet Dent 2016;115:697-702.
- 18. Mei DM, Zhao B, Xu H, Wang Y. Radiographic and clinical outcomes of rooted, platform-switched, microthreaded implants with a sandblasted, large-grid, and acid-etched surface: A 5-year prospective study. Clin Implant Dent Relat Res 2017;19:1074-81.
- 19. Al Amri MD, Abduljabbar TS. Comparison of clinical and radiographic status of platform-switched implants placed in patients with and without type 2 diabetes mellitus: a 24-month follow-up longitudinal study. Clin Oral Im- plants Res 2017;28:226-30.
- Marcello-Machado RM, Faot F, Schuster AJ, Nascimento GG, Del Bel
  Cury AA. Mini-implants and narrow diameter implants as mandibular overdenture retainers: A
  systematic review and meta-analysis of clinical and radiographic outcomes. J Oral Rehabil
  2018;45:161-83.
- 21. Al Amri MD, Kellesarian SV. Crestal bone loss around adjacent dental im- plants restored with splinted and nonsplinted fixed restorations: a systematic literature review. J Prosthodont 2017;26:495-501.
- 22. Dibart S, Warbington M, Su MF, Skobe Z. In vitro evaluation of the implant- abutment bacterial seal: the locking taper system. Int J Oral Maxillofac Im- plants 2005;20:732-7.
- 23. Stoichkov B, Kirov D. Analysis of the causes of dental implant fracture: A retrospective clinical study. Quintessence Int 2018;49:279-86.
- 24. King GN, Hermann JS, Schoolfield JD, Buser D, Cochran DL. Influence of the size of the microgap on crestal bone levels in non-submerged dental im- plants: a radiographic study in the canine mandible. J Periodontol 2002;73: 1111-7.
- 25. Blanco J, Nunez V, Aracil L, Munoz F, Ramos I. Ridge alterations following immediate implant placement in the dog: flap versus flapless surgery. J Clin Periodontol 2008;35:640-8.
- 26. Kozlovsky A, Tal H, Laufer BZ, Leshem R, Rohrer MD, Weinreb M, et al. Impact of implant overloading on the peri-implant bone in inflamed and non-inflamed peri-implant mucosa. Clin Oral Implants Res 2007;18:601-10.
- 27. Tripodi D, D'Ercole S, Iaculli F, Piattelli A, Perrotti V, Iezzi G. Degree of bacterial microleakage at the implant-abutment junction in Cone Morse tapered implants under loaded and unloaded conditions. J Appl Biomater Funct Mater 2015;13:367-71.

- Linkevicius T, Apse P, Grybauskas S, Puisys A. Influence of thin mucosal tissues on crestal bone stability around implants with platform switching: a 1- year pilot study. J Oral Maxillofac Surg 2010;68:2272-7.
- Hermann JS, Buser D, Schenk RK, Schoolfield JD, Cochran DL. Biologic width around oneand two-piece titanium implants. Clin Oral Implants Res 2001;12:559-71.
- 30. Goiato MC, dos Santos DM, Santiago JF Jr, Moreno A, Pellizzer EP. Longevity of dental implants in type IV bone: a systematic review. Int J Oral Maxillofac Surg 2014;43:1108-16.
- 31. Canullo L, Iannello G, Penarocha M, Garcia B. Impact of implant diameter on bone level changes around platform switched implants: preliminary results of 18 months follow-up a prospective randomized match-paired controlled trial. Clin Oral Implants Res 2012;23:1142-6.
- 32. Calvo-Guirado JL, Pérez-Albacete C, Aguilar-Salvatierra A, de Val Maté- Sánchez JE, Delgado-Ruiz RA, Abboud M, et al. Narrow- versus mini- implants at crestal and subcrestal bone levels. Experimental study in beagle dogs at three months. Clin Oral Investig 2015;19:1363-9.
- 33. Vohra F, Al-Kheraif AA, Almas K, Javed F. Comparison of crestal bone loss around dental implants placed in healed sites using flapped and flapless techniques: a systematic review. J Periodontol 2015;86:185-91.
- 34. Romanos GE, Javed F. Platform switching minimises crestal bone loss around dental implants: truth or myth? J Oral Rehabil 2014;41:700-8.
- 35. Kutan E, Bolukbasi N, Yildirim-Ondur E, Ozdemir T. Clinical and radio- graphic evaluation of marginal bone changes around platform-switching implants placed in crestal or subcrestal positions: a randomized controlled clinical trial. Clin Implant Dent Relat Res 2015;17:364-75.
- 36. Vela-Nebot X, Rodriguez-Ciurana X, Rodado-Alonso C, Segala-Torres M. Benefits of an implant platform modification technique to reduce crestal bone resorption. Implant Dent 2006;15:313-20.
- 37. Koutouzis T, Neiva R, Nair M, Nonhoff J, Lundgren T. Cone beam computed tomographic evaluation of implants with platform-switched Morse taper connection with the implantabutment interface at different levels in relation to the alveolar crest. Int J Oral Maxillofac Implants 2014;29:1157-63.
- Koutouzis T, Wallet S, Calderon N, Lundgren T. Bacterial colonization of the implant-abutment interface using an in vitro dynamic loading model.
   J Periodontol 2011;82:613-8.
- 39. Charalampakis G, Abrahamsson I, Carcuac O, Dahlen G, Berglundh T. Microbiota in experimental periodontitis and peri-implantitis in dogs. Clin Oral Implants Res 2014;25:1094-8.
- 40. Palaska I, Tsaousoglou P, Vouros I, Konstantinidis A, Menexes G. Influence of placement depth and abutment connection pattern on bone remodeling around 1-stage implants: a prospective randomized controlled clinical trial. Clin Oral Implants Res 2016;27:47-56.
- 41. Hamed Mortazavi; Amin Khodadousta; <u>Aida Kheiri</u>; Lida Kheiri (2021). *Bone loss-related factors in tissue and bone level dental implants: a systematic review of clinical trials.* <u>J Korean Assoc Oral Maxillofac Surg.</u> 2021 Jun 30; 47(3): 153–174.

- 42. Hamed Mortazavi; Amin Khodadoustan; Aida Kheiri; Lida.(2021). *Bone loss-related factors in tissue and bone level dental implants: a systematic review of clinical trials*. <u>J Korean Assoc Oral Maxillofac Surg.</u> 2021 Jun 30; 47(3): 153–174. Published online 2021 Jun Doi: 10.5125/jkaoms.2021.47.3.153.
- 43. Hirata, Ronaldo; Bonfante, Estevam A.; Anchieta, Rodolfo B.; Machado, Lucas S.; Freitas, Gileade; Fardin, Vinicius P.; Tovar, Nick; Coelho, Paulo G. (2016). *Reliability and failure modes of narrow implant systems. Clinical Oral Investigations, 20(7), 1505–1513.* doi:10.1007/s00784-015-1636-8
- 44. Moeintaghavi, Amir; Radvar, Mehrdad; Arab, Hamid Reza; Boostani, Hamid Reza; Ghiami, Elham (2012). Evaluation of 3- to 8-Year Treatment Outcomes and Success Rates With 6 Implant Brands in Partially Edentulous Patients. Journal of Oral Implantology, 38(S1), 441–448.doi:10.1563/AAID-JOI-D-10-00117.
- 45. L. Mahesh; G. M. Kurtzman; D. Schawrtz; S. Shukla (2015). *Residual roots as an anatomical guide for implant placement Case series with 2 year follow up...*, (), -.Doi:10.1563/aaid-joi-D-15-00101
- 46. Mehmet Ali Erdem; Burcin Karatasil; Onur Dinçer Kose; Taha Emre Kose; Erhan Çene; Serhan Aydin Aya; Abdulkadir Burak Cankaya. (2017). *The Accuracy of New and Aged Mechanical Torque Devices Employed in Five Dental Implant Systems*. <u>Biomed Res Int.</u> 2017; 2017: 8652720. Published online 2017 Nov 7. doi: 10.1155/2017/8652720.
- Mehmet Ali Erdem; Burcin Karatasli; Onur Dinçer Kose; Taha Emre Kose; Erhan Çene;
   Serhan Aydın Aya; Abdulkadir Burak Cankaya. (2017). The Accuracy of New and Aged
   Mechanical Torque Devices Employed in Five Dental Implant Systems. Biomed Res Int. 2017;
   2017: 8652720. Published online 2017 Nov7.
  - Doi: <u>10.1155/2017/8652720</u>.PMCID: PMC5697386.PMID: <u>29238725</u>.
- 48. Mahdi Kadkhodazadeh; Yaser Safi; Amir Moeintaghavi; Reza Amid; Mohammad Taghi Baghani; and Shireen Shidfar.(2019). Marginal Bone Loss Around One-Piece Implants: A 10-Year Radiological and Clinical Follow-up Evaluation. Implant Dentistry J. DOI: 10.1097/ID.0000000000000861
- 49. Tomas Linkevicius; Algirdas Puisys; Olga Svediene; Rokas Linkevicius; Laura Linkeviciene. (2015). Radiological comparison of laser- microtextured and platform-switched implants in thin mucosal biotype. Accepted 01 December 2014. To cite this article: Linkevicius T, Puisys A, Svediene O, Linkevicius R, Linkeviciene L. Radiological comparison of laser- microtextured and platform-switched implants in thin mucosal biotype. Clin. Oral Impl. Res. 00, 2015, 1–7 doi: 10.1111/clr.12544.
- 50. Roberto Rotundo; Umberto Pagliaro; Elena Bendinelli; Marco Esposito; Jacopo Buti. (2015). Long-term outcomes of soft tissue augmentation around dental implants on soft and hard tissue stability: a systematic review. Date: Accepted 12 May 2015. To cite this article: Rotundo R, Pagliaro U, Bendinelli E, Esposito M, Buti J. Long- term outcomes of soft tissue augmentation around dental implants on soft and hard tissue stability. A systematic review. Clin. Oral Impl. Res. 26 (Suppl. 11), 2015, 123–138. doi: 10.1111/clr.12629.

- 51. Daniel S. Thoma; Nadja Naenni; Elena Figuero; Christoph H. F. Hämmerle; Frank Schwarz; Ronald E. Jung; Ignacio Sanz-Sánchez.(2017). Effects of soft tissue augmentation procedures on peri-implant health or disease: A systematic review and meta-analysis. Clin Oral Impl Res. 2018;29(Suppl. 15):32–49. DOI: 10.1111/clr.13114.
- 52. Ignacio Sanz-Sánchez; Ignacio Sanz-Martín; Ana Carrillo de Albornoz; Elena Figuero; Mariano Sanz.(2018). *Biological effect of the abutment material on the stability of peri-implant marginal bone levels: A systematic review and meta-analysis. Clin Oral Impl Res.* 2018;1–21. © 2018 John Wiley & Sons A/S. | 1 Published by John Wiley & Sons Ltd. DOI: 10.1111/clr.13293.
- 53. Ronaldo Silva Cruz; Cleidiel Aparecido Araújo Lemos; Jéssica Marcela de Luna Gomes: Hiskell Francine Fernandes e Oliveira; Eduardo Piza Pellizzer; Fellippo Ramos Verri.(2020). Clinical comparison between crestal and subcrestal dental implants: A systematic review and meta-analysis. THE JOURNAL OF PROSTHETIC DENTISTRY. Copyright © 2020 by the Editorial Council for The Journal of Prosthetic Dentistry. https://doi.org/10.1016/j.prosdent.2020.11.003.
- 54. Vaishnavi Bhaskar; Hsun-Liang Chan; Mark MacEachern; Oliver D. Kripfgans. (2018). Updates on Ultrasound Research in Implant Dentistry: A Systematic Review of Potential Clinical Indications. The Authors. Published by the British Institute of Radiology. https://doi.org/10.1259/dmfr.20180076.
- 55. Manisha Herekar; Megha Sethi; Shahnawaz Mulani; Aquaviva Fernandes; Harish Kulkarni.(2014). Influence of Platform Switching on Periimplant Bone Loss: A Systematic Review and Meta-analysis. IMPLANT DENTISTRY. by Lippincott Williams & Wilkins. DOI: 10.1097/ID.000000000000000000.
- 56. Vittoria Perrotti; Daniel Zhang; Andrew Liang; Jonathan Wong; Alessandro Quaranta.(2019). The Effect of One-Abutment at One-Time on Marginal Bone Loss Around Implants Placed in Healed Bone: A Systematic Review of Human Studies. IMPLANT DENTISTRY. Wolters Kluwer Health, Inc. All rights reserved. DOI: 10.1097/ID.0000000000000931.
- 57. Saverio Cosola; Simone Marconcini; Michela Boccuzzi; Giovanni Battista Menchini Fabris; Ugo Covani; Miguel Peñarrocha-Diago; David Peñarrocha-Oltra. (2020). *Radiological Outcomes of Bone-Level and Tissue-Level Dental Implants: Systematic Review. Int. J. Environ. Res. Public Health* 2020, *17*, 6920; doi:10.3390/ijerph17186920.
- 58. Cosyn J, Hooghe N, De Bruyn H. A systematic review on the frequency of advanced recession following single immediate implant treatment. J Clin Periodontol 2012; 39: 582–589. doi: 10.1111/j.1600-051X.2012.01888.x.
- 59. Felipe Cáceres' Cristian Troncoso; Ramón Silva; Nelson Pinto. (2020). Effects of osseodensification protocol on insertion, removal torques, and resonance frequency analysis of BioHorizons® conical implants. An ex vivo study. 2212-4268/ © 2020 Craniofacial Research Foundation. Published by Elsevier B.V. All rights reserved. https://doi.org/10.1016/j.jobcr.2020.08.019.

- 60. Mohammad D. Al Amri. (2016). *Crestal bone loss around submerged and nonsubmerged dental implants: A systematic review*. THE JOURNAL OF PROSTHETIC DENTISTRY. Prosthet Dent. 2016 May;115(5):564-570.e1. Doi: 10.1016/j.prosdent.2015.11.002.
- 61. Zhaozhao Chen; Cho-Ying Lin; Junying Li; Hom-Lay Wang; Haiyang. (2019). *Influence of abutment height on peri-implant marginal bone loss: A systematic review and meta-analysis.* J Prosthet Dent. 2019 Jul;122(1):14-21.e2. Doi: 10.1016/j.prosdent.2018.10.003.
- 62. Naser Sargolzaie; Sarah Samizade; Hamidreza Arab; Habibollah Ghanbari; Leila Khodadadifard; Amin KhajavI. (2019). *The evaluation of implant stability measured by resonance frequency analysis in different bone types*. Korean Assoc Oral Maxillofac Surg. 2019 Feb;45(1):29-33. Doi: 10.5125/jkaoms.2019.45.1.29.Epub 2019 Feb 26.
- 63. Michael R Norton; Mikael Astrom. (2020). The Influence of Implant Surface on Maintenance of Marginal Bone Levels for Three Premium Implant Brands: A Systematic Review and Meta-analysis. Int J Oral Maxillofac Implants. Nov/Dec 2020;35(6):1099-1111.Doi: 10.11607/jomi.8393.
- 64. Kirsten W. Slagter; Laurens den Hartog; Nicolaas A. BakkeR; Arjan Vissink; Henny J.A. Meijer; Gerry M. Raghoebar. (2014). *Immediate placement of dental implants in the esthetic zone: a systematic review and pooled analysis*. J Periodontol 2014 Jul;85(7):e241-50.Doi: 10.1902/jop.2014.130632. Epub 2014 Feb 6.
- 65. Zhaozhao Chen; Yujiao Zhang; Junying; Hom-lay Wang; Haiyang. (2017). *Influence of Laser-Microtextured Surface Collar on Marginal Bone Loss and Peri-Implant Soft Tissue Response: A Systematic Review and Meta-Analysis*. J Periodontol. 2017 Jul;88(7):651-662.Doi: 10.1902/jop.2017.160805. Epub 2017 Mar 17.
- 66. Seyed Hossein Bassir; Karim El Kholy; Chia-Yu Chen; Kyu Ha Lee; Giuseppe Intini. (2019). Outcome of early dental implant placement versus other dental implant placement protocols: A systematic review and meta-analysis. J Periodontol. 2019 May;90(5):493-506. Doi: 10.1002/JPER.18-0338. Epub 2018 Dec 5.
- 67. Lorenzo Tavelli; Shayan Barootchi; Gustavo Avila-Ortiz†; Istvan Urban; William V. Giannobile; Hom-Lay Wang. (2021). Peri-implant Soft Tissue Phenotype Modification and its Impact on Peri-Implant Health: A Systematic Review and Network Meta-Analysis. J Periodontol. 2021 Jan;92(1):21-44. Doi: 10.1002/JPER.19-0716. Epub 2020 Aug 9.
- 68. Mahdi Kadkhodazadeh; Reza Amid; Anahita MoscowchI.(2022). *Impact of collar laser microtexturing on peri-implant health and disease: a retrospective clinical study*. Clin Oral Investig. 2022 Feb;26(2):1637-1645.Doi: 10.1007/s00784-021-04136-8. Epub 2021 Aug 16.
- 69. Hilario Pellicer-Chover; María Peñarrocha-Diago; David Peñarrocha-Oltra; Sonia Gomar-Vercher; Rubén Agustín-Panadero; Miguel Peñarrocha-Diago. (2016). *Impact of crestal and subcrestal implant placement in peri-implant bone: A prospective comparative study.* Med Oral Patol Oral Cir Bucal. 2016 Jan 1;21 (1):e103-10. Crestal and subcrestal implant placement. *Journal section: Oral Surgery Publication Types: Research Doi:10.4317/medoral.20747 http://dx.doi.org/doi:10.4317/medoral.20747*.

- 70. Cristina Valles; Xavier Rodríguez-Ciurana; Marco Clementini; Mariana Baglivo; Blanca Paniagua; Jose Nart.(2018). *Influence of subcrestal implant placement compared with equicrestal position on the peri-implant hard and soft tissues around platform-switched implants: a systematic review and meta-analysis*. Clinical Oral Investigations. Published online: 08 January 2018. <a href="https://doi.org/10.1007/s00784-017-2301-1">https://doi.org/10.1007/s00784-017-2301-1</a>.
- 71. De Medeiros FCFL, Kudo GAH, Leme BG, Saraiva PP, Verri FR, Honório HM, Pellizzer EP, Santiago Junior JF. *Dental implants in patients with osteoporosis: a systematic review with meta-analysis. Int J Oral Maxillofac Surg* 2018; 47: 480-491. pii: S0901- 5027(17)31484-4. doi: 10.1016/j.ijom.2017.05.021.[Epub ahead ofprint] Review. PubMed PMID: 28651805.
- 72. Al Amri MD, Al-Johany SS, Al Baker AM, Al Rifaiy MQ, Abduljabbar TS, Al-Kheraif AA (2016) Soft tissue changes and crestal bone loss around platform-switched implants placed at crest- al and subcrestal levels: 36-month results from a prospective split- mouth clinical trial. Clin Oral Implants Res 28(11):1342–1347. https://doi.org/10.1111/clr.12990
- 73. Gale NK, Heath G, Cameron E, Rashid S, Redwood S. Using the framework method for the analysis of qualitative data in multi-disciplinary health research. BMC Medical Research Methodology. 2013 Dec 18;13(1):117.
- 74. Casagrande A, Fabris F, Girometti R. Beyond kappa: an informational index for diagnostic agreement in dichotomous and multivalue ordered-categorical ratings. Medical & biological engineering & computing. 2020 Dec;58(12):3089–99.